CLINICAL TRIAL: NCT03707288
Title: The Prevalence of Neck and Low Back Pain in Medical Students at The University of the West Indies, Mona, Jamaica
Brief Title: Neck and Low Back Pain in Medical Students at The University of the West Indies, Mona, Jamaica
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Collaborators: The University of The West Indies, Mona (Unknown)
Responsible Party: Principal Investigator, Paula Dawson, MBBS, Head, Physical Medicine and Rehabilitation. Principal Investigator, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ECP 248, 13/14
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Back Pain; Low Back Pain; Neck Pain; Neck Pain Musculoskeletal; Lower Back Pain; Spine Health; Musculoskeletal Pain; Musculoskeletal Pain Disorder
Keywords: lower back pain; low back pain; neck pain; neck and back pain; spine health; medical students; university students; musculoskeletal pain
MeSH Terms: conditions — Back Pain; Low Back Pain; Neck Pain; Musculoskeletal Pain; Collagen Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Control (Group A) (Other): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group A will not be given any exercise programs over an eight (8) week period after which time, participants will be reassessed using the CMDQ and NRS, as well as a Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, without having received any intervention.
  Interventions: Behavioral: Clinical Control Group (Group A)
- Spine Exercise Program (Group B) (Other): All participants will complete the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess the frequency, discomfort and interference with work due to musculoskeletal pain; the Numeric Rating Scale (NRS) to assess for perceived pain; as well as Questionnaire A to assess their knowledge, attitude and practice towards musculoskeletal problems of neck or low back pain. Participants who are found to have neck or low back pain will be randomised into two (2) groups: a clinical control group (Group A) and an intervention group (Group B). Group B will be given a standardised spine exercise program over an eight (8) week period, after which time they will be reassessed using the CMDQ and NRS, as well as Questionnaire B to evaluate for changes in their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, having received the intervention.
  Interventions: Behavioral: Spine Exercise Program (Group B)

INTERVENTIONS:
Behavioral: Clinical Control Group (Group A) — The participants who reported the presence of neck or low back pain and were assigned to the clinical control group (Group A) after randomisation will not receive the intervention of an exercise program. The interventional group (Group B) will be asked to keep the standardised exercise program confidential and not share with the control group (Group A). After eight (8) weeks, Group A participants will receive: the Cornell Musculoskeletal Discomfort Questionnaires (CMDQ) to assess for changes in the frequency, discomfort and interference with work due to musculoskeletal pain; a Questionnaire B, to ascertain any changes in their pain level using the Numeric Rating Scale (NRS); as well as their knowledge, attitude and practice towards musculoskeletal problems of the neck and low back pain, without having received any intervention.
  Arms: Clinical Control (Group A)
Behavioral: Spine Exercise Program (Group B) — The standardised spine exercise program will be provided in a handout and given only to the intervention group (Group B), and will include simple basic neck or low back exercises to be done three (3) times per week, as well as brief stretching exercises, to be done during periods of sitting for greater than sixty (60) minutes. The selected participants will be asked to comply with instructions on the handout. Participants who experience worsening of their symptoms, or who develop new symptoms will be assessed as having an adverse outcome and will be withdrawn from the study.
  Arms: Spine Exercise Program (Group B)

SUMMARY:
The purpose of this study is to identify the prevalence of neck and low back pain in medical students enrolled at the University of the West Indies, Mona; to assess their knowledge, attitude and practice of good spine health and to determine the outcome of a standardised spine exercise program on medical students experiencing neck and low back pain, using a prospective randomised control design.

DETAILED DESCRIPTION:
There is a surfeit of literature on musculoskeletal pain especially that of neck and low back pain, which are commonly associated with lifestyle practices including varied occupations that affect individuals of all ages.

Medical students in the clinical years of training are more likely to be involved in prolonged and strenuous activities such as standing during ward rounds, bending forward to examine patients and occasionally engaging in manual handling of patients. During the early phase of preclinical training, medical students primarily sit for extended periods in lectures, use computers or tablets, or study in the library while completing assignments. These practices may all contribute to the increased risk of developing neck and low back pain among other musculoskeletal problems, especially in instances where the strength and stability of the spine is not maintained and safe spine precautions are not taken.

To the researcher's knowledge, there is no published study in Jamaica, or in the wider Caribbean, which looks at the prevalence of musculoskeletal pain -- specifically neck and low back pain in medical students. This study aims to determine the prevalence of neck and low back pain in medical students at the University of the West Indies (UWI), Mona, as well as to assess their knowledge, attitude and practice toward good spine health in preventing neck and low back pain.

Using a prospective randomised control study model for students experiencing neck and low back pain, this study will evaluate the outcome of a standardised spine exercise program in participants over an eight (8) week period. These participants will be randomly assigned to the clinical control group (Group A), which will receive no intervention, or the intervention group (Group B), which will follow a standardised spine exercise program over the stipulated period. Data will be collected using Questionnaires A and B, the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), and the Numeric Rating Scale (NRS). The outcomes of both groups will then be compared to determine the program's effectiveness in reducing discomfort and promoting better knowledge, attitude and practice towards spine health among medical students.

The identity of all participants will be protected and will only be identified by an assigned study number. Basic demographic information, presenting complaints and outcome information will be obtained for the purposes of the study. All data will be managed securely using REDCap, a password-protected, web-based platform compliant with national data protection standards. Data exported for analysis will be handled using SPSS software, ensuring confidentiality is maintained throughout. All records will be securely destroyed three years after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. All students enrolled in the medical program at the University of the West Indies, Mona Campus, Jamaica during the period October 1, 2018 to January 2, 2026.
2. Individuals who express a willingness to consent to the study.
3. Individuals who express a willingness to adhere to the standardised exercise program for the stipulated period.

Exclusion Criteria:

1. Individuals with a history of having spine surgery.
2. Individuals who were previously diagnosed with spine pathology and currently receiving rehabilitation therapy.
3. Individuals who express an unwillingness to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender males and females
Enrollment: 1000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | From enrollment to the end of treatment at eight (8) weeks
  The Cornell Musculoskeletal Discomfort Questionnaire measures the frequency, discomfort and interference with work due to musculoskeletal pain, as reported by participants. The individually reported frequency score is then multiplied by the discomfort score and by the interference score to determine overall severity of pain experienced. This tallied score is then classified by severity into: no discomfort (0), mild (1 to 4.5), moderate (5 to 14), severe (15 - 45) and very severe (45 or higher). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their reported scores.

SECONDARY OUTCOMES:
Knowledge, Attitude and Practice towards Musculoskeletal Problems of Neck and Low back Pain (Questionnaire A) | Done at the time of enrollment (Baseline)
  Questionnaire A is a self-administered general questionnaire used to evaluate knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in Knowledge, Attitude and Practice Towards Musculoskeletal Problems of Neck and Low Back Pain (Questionnaire B) | From Enrollment to the end of treatment at 8 weeks
  Questionnaire B is a self-administered general questionnaire used to evaluate changes in knowledge, attitude and practice towards musculoskeletal problems of neck and low back pain.
Change from Baseline in the Numeric Rating Scale (NRS) | From Enrollment to the end of treatment at 8 weeks
  The Numeric Rating Scale is a reliable and valid, unidimensional 11-point scale used for patient self-reporting of perceived pain. Its scale uses integers which range from zero (0) to ten (10), where 0 represents no pain, and 10 represents the worst imaginable pain. This is then categorised into mild (1-3), moderate (4-6), and severe (7-10). All participants will complete this assessment upon enrollment, as well as after an eight (8) week period of treatment, to evaluate any changes in their perceived pain. This scale is from public domains and as such, permission for its use is not required.

CONTACTS AND LOCATIONS:
Overall Officials: Paula U. A. Dawson, MBBS, Diplomate ABPMR, Principal Investigator — Division of Physical Medicine and Rehabilitation, Faculty of Medical Sciences, The University of the West Indies, Mona, Jamaica.
Locations (2):
- Jamaica (2):
  - Faculty of Medical Sciences Teaching and Research Complex,The University of the West Indies, University Hospital of the West Indies, Kingston, Kingston
  - Faculty of Medical Sciences Teaching and Research Complex, University of The West Indies-Mona Campus, Kingston

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ehrlich GE. Low back pain. Bull World Health Organ. 2003;81(9):671-6. Epub 2003 Nov 14. PMID 14710509
- [Background] Punnett L, Pruss-Utun A, Nelson DI, Fingerhut MA, Leigh J, Tak S, Phillips S. Estimating the global burden of low back pain attributable to combined occupational exposures. Am J Ind Med. 2005 Dec;48(6):459-69. doi: 10.1002/ajim.20232. PMID 16299708
- [Background] Lis AM, Black KM, Korn H, Nordin M. Association between sitting and occupational LBP. Eur Spine J. 2007 Feb;16(2):283-98. doi: 10.1007/s00586-006-0143-7. Epub 2006 May 31. PMID 16736200
- [Background] Smith DR, Wei N, Ishitake T, Wang RS. Musculoskeletal disorders among Chinese medical students. Kurume Med J. 2005;52(4):139-46. doi: 10.2739/kurumemedj.52.139. PMID 16639985
- [Background] Falavigna A, Teles AR, Mazzocchin T, de Braga GL, Kleber FD, Barreto F, Santin JT, Barazzetti D, Lazzaretti L, Steiner B, Beckenkamp NL. Increased prevalence of low back pain among physiotherapy students compared to medical students. Eur Spine J. 2011 Mar;20(3):500-5. doi: 10.1007/s00586-010-1646-9. Epub 2010 Dec 7. PMID 21136121
- [Background] Alshagga MA, Nimer AR, Yan LP, Ibrahim IA, Al-Ghamdi SS, Radman Al-Dubai SA. Prevalence and factors associated with neck, shoulder and low back pains among medical students in a Malaysian Medical College. BMC Res Notes. 2013 Jul 1;6:244. doi: 10.1186/1756-0500-6-244. PMID 23815853
- [Background] Smith DR, Leggat PA. Musculoskeletal disorders among rural Australian nursing students. Aust J Rural Health. 2004 Dec;12(6):241-5. doi: 10.1111/j.1440-1854.2004.00620.x. PMID 15615575
- [Background] Lorusso A, Vimercati L, L'abbate N. Musculoskeletal complaints among Italian X-ray technology students: a cross-sectional questionnaire survey. BMC Res Notes. 2010 Apr 24;3:114. doi: 10.1186/1756-0500-3-114. PMID 20416101
- [Background] Smith DR, Leggat PA, Walsh LJ. Workplace hazards among Australian dental students. Aust Dent J. 2009 Jun;54(2):186-8. doi: 10.1111/j.1834-7819.2009.01116_8.x. No abstract available. PMID 19473172
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Mandel JH, Lohman W. Low back pain in nurses: the relative importance of medical history, work factors, exercise, and demographics. Res Nurs Health. 1987 Jun;10(3):165-70. doi: 10.1002/nur.4770100308. PMID 2954190
- [Background] Ariens GA, van Mechelen W, Bongers PM, Bouter LM, van der Wal G. Physical risk factors for neck pain. Scand J Work Environ Health. 2000 Feb;26(1):7-19. doi: 10.5271/sjweh.504. PMID 10744172